CLINICAL TRIAL: NCT06571032
Title: Evaluation of Electroencephalography in the Management of Neuroelectric Stimulation in Patients With Severe Traumatic Brain Injuries: A Prospective Study
Brief Title: Electroencephalography in the Management of Neuroelectric Stimulation in Patients With Severe Traumatic Brain Injuries
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Junfeng Feng, Director of Brain Injury Center, RenJi Hospital
Other Study IDs: LY2024-007
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Brain Injuries
Keywords: Electroencephalography; Severe traumatic brain injuries
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Consicousness improved group: After receiving neuroelectrial stimulation, the patients with severe TBI have the consciousness improvement (CRS-R score is higher than before).
- Consicousness unimproved group: After receiving neuroelectrial stimulation, the patients with severe TBI have no consciousness improvement (CRS-R score remains the same as before).

SUMMARY:
The goal of this observational retrospective study is to evaluate the electroencephalography (EEG)'s poficiency in the treatment of neuroelectric stimulation in patients with severe traumatic brain injuries (TBI).

The main questions it aims to answer are:

1. Whether EEG of patients with severe TBI will change after they receiving neuroelectrial stimulation? If yes, how does it change?
2. How can EEG be used to evaluate the condition of patients with severe TBI?

ELIGIBILITY:
Inclusion Criteria:

* 7 days after severe traumatic brain injuries (GCS score 3-8);
* Over 18 years old, regardless of gender;
* The patient's legal representative is informed and voluntarily signs the consent form.

Exclusion Criteria:

* Unstable vital signs;
* History of mental disorders or neurodegenerative diseases;
* Uncontrolled epilepsy;
* Severe arrhythmias or patients with implanted cardiac pacemakers;
* Various conditions that interfere with scalp EEG collection;
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients have severe TBI and receive neuroelectral stimulation.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-08-14 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
CRS-R scores 6 months after the patient's discharge | 6 months
  Using the COMA RECOVERY SCALE-REVISED (CRS-R) to evaluate the condition of the patient 6 months after discharge and the effectiveness of neuroelectrial stimulation. The minimum and maximum values of CRS-R is 0 and 23 and higher scores mean a better outcome.

SECONDARY OUTCOMES:
CRS-R scores during hospitalization | 3 months
  Using the COMA RECOVERY SCALE-REVISED (CRS-R) to evaluate the condition of the patient during hospitalization and the effectiveness of neuroelectrial stimulation. The minimum and maximum values of CRS-R is 0 and 23 and higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Junfeng Feng, Ph.D., Principal Investigator — RenJi Hospital
Locations (1):
- Brain Injury Center, Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided